CLINICAL TRIAL: NCT04302077
Title: Patient Satisfaction With Virtual Post Operative Visits: Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-01949
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemedicine Post Op (Active Comparator): Patients with an even-ending medical record number (0,2,4,6,8) will be randomized to virtual visit/telemedicine. This will be done by using Epic and MyChart-integrated telemedicine functionality for video visits with the Principal Investigator's patients. This is considered standard of care.
  Interventions: Other: virtual doctor visit
- In-Office Post Op (Active Comparator): Patients with an odd-ending medical record number (1,3,5,7,9) will be randomized to the office visit.
  Interventions: Other: Standard care doctor's visit

INTERVENTIONS:
Other: virtual doctor visit — interactive live-video feed at home through EPIC
  Arms: Telemedicine Post Op
Other: Standard care doctor's visit — In person visit as per standard of care
  Arms: In-Office Post Op

SUMMARY:
This is a prospective, randomized study designed to evaluate the effects of different initial postoperative follow-up modalities. Given the nature of the study, it is not possible for either the surgeons or the subjects to be blinded. Patients will be assigned to either group based on the last digit of their medical record number (MRN). Patients with an even-ending medical record number will be randomized to virtual visit/telemedicine, while patients with an odd-ending medical record number will be randomized to the office visit.

DETAILED DESCRIPTION:
This study aims to evaluate the differences between two forms of postoperative follow-up with respect to patient satisfaction. The primary outcome will be patient satisfaction with their surgeon and with their overall experience. Following their second postoperative visit, the subjects will complete one electronic survey. The survey is designed to assess subject's overall satisfaction and satisfaction with their surgery. This survey is standardized and will be used by both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing arthroscopic hip surgery

Exclusion Criteria:

* Age < 18 years old or Age > 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction | 3 month follow up visit
  Participant satisfaction will be measured by a electronic survey . At the conclusion of the in-person or virtual visit, participants will be provided instructions how to access the survey questions through the QR code if in-person and through a secure link if at home via telemedicine through EPIC.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to jordan.fried@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.